CLINICAL TRIAL: NCT04077970
Title: Evaluation of Implantation and Clinical Pregnancy After Intrauterine Flushing of Infertile Patients With Follicular Fluid Plus Granulosa Cells- Randomized Controlled Trial
Brief Title: Intrauterine Flushing With Follicular Fluid Plus Granulosa Cells
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Infertility-Uterine flushing
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Follicular Fluid; Granulosa Cell; Embryo Implantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrauterine flushing follicular fluid (Experimental): Women underwent intrauterine flushing with follicular fluid plus granulosa cells
  Interventions: Biological: Intrauterine flushing of follicular fluid with granulosa cells
- Without intrauterine flushing with follicular fluid (No Intervention): Women without intrauterine flushing with follicular fluid

INTERVENTIONS:
Biological: Intrauterine flushing of follicular fluid with granulosa cells — All patients in case and control groups will receive agonist and antagonist protocol. Ovarian stimulation will be carried out when pituitary desensitization is achieved and is continued until the day of hCG administration. COCs aspiration will be performed 34-36h after hCG injection. Clear Follicular Fluids (without blood cells) which contain COCs will be used. Endometrial flushing after oocyte retrieval with 2 ml of clear FF plus granulose cells will be performed by an IUI catheter. The control group included 70 women who would not have FF endometrial flushing. In both groups, embryo transfer will be carried out 2-3 days later. Luteal phase support will be started the day after ovum pick up by the vaginal administration of progesterone daily for 16 days and will continued for up to12 weeks if pregnancy occurred. Pregnancy was diagnosed by measurement of β-hCG level and later was confirmed by Transvaginal sonography.
  Arms: Intrauterine flushing follicular fluid

SUMMARY:
One hundred forty patients with male factor infertility are randomized into two groups. In the study group, flushing the endometrial cavity with 2ml of clear follicular fluid with granulose cells will be performed using an IUI catheter after ovum pick-up While in the control group, no flushing of the endometrial cavity with FF is done. The implantation rates and pregnancy rates in both groups will be assessed.

DETAILED DESCRIPTION:
This study is a randomized clinical trial to investigate implantation rate and clinical pregnancy after intrauterine flushing of infertile patients with follicular fluid plus granulosa cells - Randomized controlled trials. The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute and all participants provide informed consent.

The main objective of this study is evaluation of implantation rate and clinical pregnancy after flushing of uterine in infertile patients with follicular fluid plus granulosa cells in IVF/ ICSI cycles.

Material and methods: In a randomized clinical trial, 140 patients with Male factor infertility referring to infertility clinic of Royan Institute, Iran, who received ovarian stimulation with antagonist and agonist protocol, will be randomly assigned to two groups: in case group, if the follicular fluid of two clear dominant follicles contain at least 2 COC, after removal of the COCs, follicular fluid will be collected Endometrial cavity flushing with 2 ml of follicular fluid will be performed by IUI caterer. In control group only catheterization of uterine cavity will be performed. Primary outcome is comparison of implantation rate between case and control group. Secondly outcome is assessment of clinical pregnancy rate in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Normal Hormonal profile (FSH, LH, AMH) and normal AFC
2. Normal ovarian reserve
3. Age 20-38 years
4. Regular menstrual cycle
5. IVF / ICSI or IVF or ICSI cycles with agonist and antagonist protocol
6. Existence of at least 2 oocytes in dominant follicular fluids

Exclusion Criteria:

1. Presence of Endometriosis and Endometrioma
2. Hydrosalpinx
3. OHSS (Ovarian Hyper Stimulating Syndrome)
4. Tubal factor infertility
5. Male factor infertility with azoospermia
6. Low/Poor Response
7. Myoma with a compression effect or submocusa myometrium
8. Intra mural or subserouse Myoma > 5cm
9. Presence of untreated Thyroid, Diabetic and Hepatitis diseases, vaginal infection.
10. Endometrial tuberculosis
11. The follicular fluid which contains any oocyte or contaminated with blood will be discarded

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Implantation rates | Day 35-42 post ovum pick-up (OPU) (34-36 hours post recombinant human choriogonadotropin day [approximately 28 days])
  Implantation rate was measured as the number of gestational sacs observed, divided by the number of embryos transferred

SECONDARY OUTCOMES:
Clinical pregnancy rate | 4-6 weeks after embryo transfer
  The observation of gestational sac on ultrasound examination two-three weeks after positive serum βhCG

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Hafezi, Study Chair — Department of Endocrinology and Female Infertility
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Hosseini E, Aghajanpour S, Chekini Z, Zameni N, Zolfaghary Z, Aflatoonian R, Hafezi M. An Approach to Improve Endometrial Receptivity: Is It Beneficial to Flush The Uterine Cavity with Follicular Fluid and Granulosa Cells? A Phase III Randomised Clinical Trial. Int J Fertil Steril. 2024 Jul 13;18(Suppl 1):22-29. doi: 10.22074/ijfs.2023.2000897.1461. PMID 39033367